CLINICAL TRIAL: NCT05526339
Title: High-Flow Nasal Oxygenation Combined With Nasopharyngeal Airway Reduces The Incidence Of Hypoxia During Gastrointestinal Endoscopy Sedated With Propofol In Obese Patients: A Prospective, Randomized Clinical Trial
Brief Title: HFNO Combined With NPA Reduces Hypoxia During Sedated Gastrointestinal Endoscopy In Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Second Affiliated Hospital of Soochow University (Other); Dushu Lake Hospital Affiliated to Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LY2022-018-A
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer; Gastric Ulcer; Intestinal Cancer; Intestinal Polyps
Keywords: High-flow nasal oxygenation; Gastrointestinal endoscopy; Hypoxia
MeSH Terms: conditions — Stomach Neoplasms; Stomach Ulcer; Intestinal Neoplasms; Intestinal Polyps; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal oxygenation combined with nasopharyngeal airway (Experimental): High-flow nasal oxygenation combined with nasopharyngeal airway was used in obese patients who are scheduled to undergo gastrointestinal endoscopy procedures sedated with propofol.
  Interventions: Device: High-flow nasal oxygenation combined with nasopharyngeal airway
- Regular nasal cannula combined with nasopharyngeal airway (Active Comparator): Regular nasal cannula combined with nasopharyngeal airway was used in obese patients who are scheduled to undergo gastrointestinal endoscopy procedures sedated with propofol.
  Interventions: Device: Regular nasal cannula combined with nasopharyngeal airway

INTERVENTIONS:
Device: High-flow nasal oxygenation combined with nasopharyngeal airway — The patients receive an oxygen flow of 30 L/min for preoxygenation with a high-flow oxygenation device before losing of conscious. At the time of the abolition of the eyelash reflex, the gas flow was increased to 60 L/min with an inspired oxygen fraction 100% and the nasopharyngeal airway was placed.
  Arms: High-flow nasal oxygenation combined with nasopharyngeal airway
Device: Regular nasal cannula combined with nasopharyngeal airway — The patients receive an oxygen flow of 6 L/min for preoxygenation with a regular nasal cannula until the end of procedure. At the time of abolition of the eyelash reflex, the nasopharyngeal airway was placed.
  Arms: Regular nasal cannula combined with nasopharyngeal airway

SUMMARY:
Obesity is associated with adverse airway events including desaturation during deep sedation. Previous studies have suggested that high-flow nasal oxygenation may be superior to regular (low-flow) nasal cannula for prevention of hypoxia during Sedated Gastrointestinal Endoscopy in non-obesity patients. The prerequisite of high-flow nasal oxygenation is keeping airway patency. Our pervious study demonstrated that nasopharyngeal airway has the similar efficacy of jaw-lift. In present study we aimed to determine whether high-flow nasal oxygenation combined with nasopharyngeal airway could reduce the incidence of hypoxia during Sedated Gastrointestinal Endoscopy in obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving selective combined upper intestinal and lower intestinal endoscopy procedure under deep sedation.
2. Age ranging from 19 to 80, both male and female
3. Obese patients，BMI ≥ 28kg/m^2
4. ASA I~III
5. Patients should clearly understand and voluntarily participate in the study, with signed informed consent.

Exclusion Criteria:

1. Patients with acute respiratory infection in the last 2 weeks
2. Patients with nasal congestion, epistaxis, recent nasal trauma, recent nasal surgery
3. hypoxia, defined as oxygen saturation measured by pulse oximetry (SpO2) ≤ 95% before preoxygenation.
4. Common advanced gastrointestinal endoscopy procedures meeting eligibility criteria included cholangiopancreatography, endoscopic ultrasound procedures, endoscopic mucosal resection and endoscopic retrograde cholangiopancreatography (ERCP) procedures.
5. coagulation disorders or platelets < 100*10^9/L
6. Have serious heart diseases such as severe arrhythmia, heart failure, Adams Stokes Disease, unstable angina pectoris, myocardial infarction in the last 6 months, history of tachycardia / bradycardia requiring medical treatment, third degree atrioventricular block or QTC interval ≥ 450ms (corrected according to fridericia's formula), or exercise tolerance < 4mets
7. Allergy to eggs, soy products, opioids and other drugs, propofol, etc.
8. Participated in other clinical trials as a subject within 3 months
9. Patients with brain injury, possible convulsion, myoclonus, intracranial hypertension, cerebral aneurysm, cerebrovascular accident history, schizophrenia, intellectual disability, mania, psychosis, long-term use of psychotropic drugs, drug addiction, cognitive dysfunction history, etc.
10. Emergency procedure
11. Pregnant or breast-feeding women
12. Patients having procedures with planned tracheal intubation or laryngeal mask
13. Investigator considers the patients are inappropriate to participate in this trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Hypoxia refers to 75%≤SpO2<90%,<60S

SECONDARY OUTCOMES:
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Severe hypoxia refers to SpO2<75% lasting for any time, or 75%≤SpO2<90%, ≥60s
The incidence of subclinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Subclinical respiratory depression refers to 90%≤ SpO2<95%
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Principal Investigator — RenJi Hospital
Locations (2):
- China (2):
  - Dushu Lake Hospital Affiliated to Soochow University, Suzhou, Jiangsu
  - Second Hospital Affiliated to Soochow University, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No